CLINICAL TRIAL: NCT06231056
Title: Probiotic Therapy in Pregnancy for the Reduction of Streptococcus Agalactiae Positivity and the Frequency of PROM, pPROM and Preterm Birth
Brief Title: Probiotic Supplementation as Prophylactic for Group B β-hemolytic Streptococcus (GBS) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LUMHS/iNatal/20.01.2024
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Genitourinary; Infection, Complicating Pregnancy
MeSH Terms: conditions — Infections; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Probiotic supplement group
Masking Description: Control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplement group (Experimental): Participants in this group received probiotic iNatal® (Enterococcus faecium L3, Bifidobacterium animalis subsp. lactis BB-12, Lactococcus lactis SP38, Lacticaseibacillus casei R0215) - dosage 1 sachet per day, during the 24-36 weeks of their gestation period.
  Interventions: Dietary Supplement: Probiotic iNatal®
- Control group (No Intervention): No probiotic supplementation. Participants in this group did not received probiotic iNatal® during 24-36 weeks of their gestation period.

INTERVENTIONS:
Dietary Supplement: Probiotic iNatal® — iNatal® (Enterococcus faecium L3, Bifidobacterium animalis subsp. lactis BB-12, Lactococcus lactis SP38, Lacticaseibacillus casei R0215)
  Arms: Probiotic supplement group

SUMMARY:
Streptococcus agalactiae, a Group B β-hemolytic streptococcus (GBS), is the leading cause of severe neonatal infection in developed countries. There is growing scientific interest in probiotic supplementation in pregnancy as possible prophylaxis for GBS infections and urine culture positivity.

DETAILED DESCRIPTION:
There is strong scientific evidence that supports the correlation between bacterial vaginosis (BV), a term used to define a change in the vaginal ecosystem, and spontaneous preterm birth. Antibiotic treatments are recommended to counteract both the presence of S. agalactiae and the onset of BV. The latter, however, are not without risks, as they can in turn cause alterations in the vaginal microbiota and is associated with an increased risk of miscarriage.

Recent research have shown that probiotic treatment can help reduc the risk of preterm birth and positivity of Group B β-hemolytic streptococcus (GBS) infection.

The present study aimed to assess the efficacy and safety of a probiotic iNatal® (probiotic mixture containing 10 ml CFU of Enterococcus faecium L3, 3 billion CFU of Bifidobacterium animalis subsp. lactis BB-12, 3 billion CFU of Lactococcus lactis SP38, 3 billion CFU of Lacticaseibacillus casei R0215) in pregnant wemen in 24 to 36 weeks of gestation as prophylaxis of GBS infections and urine culture positivity.

This was a retrospective, observational, controlled and single centre study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in 24-36 weeks of gestation period
* History of recurrent genitourinary and/or intestinal problems

Exclusion Criteria:

* Presence of neurological condition
* History of cardiovascular disease
* History of pulmonary disease
* History of renal disease
* Cancer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is only applicable in pregnant female.
Enrollment: 250 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Bacteriological assessment | 12 weeks
  Control of bacteriuria by urine culture (number of participants)
Bacteriological assessment | 12 weeks
  Incidencce of Group B β-hemolytic streptococcus (GBS) infection positivity investigation by vaginal and/or rectal swab
Clinical assessments at the end of pregnancy | 12 weeks
  Incidence of Prelabor rupture of membranes (PROM)
Clinical assessments at the end of pregnancy | 12 weeks
  Incidence of Preterm PROM (PPROM)
Clinical assessments at the end of pregnancy | 12 weeks
  Incidence of Preterm birth
clinical assessments at the end of pregnancy | 12 weeks
  Rate of natural or caesarean section mode
Clinical assessments at the end of pregnancy | 12 weeks
  Incidence of induction of child birth

SECONDARY OUTCOMES:
Rate of incidence of side effects | 12 weeks
  Number of participants presenting any side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology PERUGIA HOSPITAL, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No